CLINICAL TRIAL: NCT05078541
Title: A Safety and Feasibility Trial of Ultrasound Guided Radiofrequency Ablation of Parotid Warthin's Tumor
Brief Title: Radiofrequency Ablation for Warthin's Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, David Yeung, Resident, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2021.412
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Safety and Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA Warthins Tumor Group (Experimental): Group of patients who will under RFA for Warthin's tumor.
  Interventions: Procedure: Ultrasound-guided Radiofrequency Ablation of Parotid Warthin's Tumor

INTERVENTIONS:
Procedure: Ultrasound-guided Radiofrequency Ablation of Parotid Warthin's Tumor — The Procedure
  1. Injection of local subcutaneous and pericapsular anaesthesia
  2. Needle radiofrequency ablation under ultrasound guidance
  3. Patients should communicate with operating surgeon upon excessive heat or pain
  4. The procedure usually lasts 30-45 minutes

SUMMARY:
This study is a safety and feasibility study to determine if ultrasound guided radiofrequency ablation of parotid Warthin's tumor under local anesthesia is a safe and effective procedure compared to Parotidectomy while using less resources.

DETAILED DESCRIPTION:
Radiofrequency ablation is minimally invasive and is used in benign disease, including thyroid nodules, head and neck nodules, and vascular malformations, as well as some malignant tumors. For patients unable to or unwilling to undergo surgical resection, real-time ultrasound guided radiofrequency ablation for parotid Warthin's Tumor would be a further option besides observation alone.

Twenty patients with Warthin's tumor from the ENT Head and Neck Surgery out-patient clinic at Prince of Wales Hospital will be recruited. The patient will first be asked if they wanted intervention for their condition of Warthin's Tumor. Parotidectomy will first be offered. If the patient opted for intervention but declines parotidectomy, then ultrasound guided RFA will be offered.

The 2019 - 2020 Parotidectomy for Warthin's tumor internal audit will be used as a historical comparison to the ultrasound guided RFA group.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Ultrasound scan findings:

   1. Tumor size 2cm-5cm
   2. Tumor located in superficial lobe of parotid gland with epicenter in Parotid tail
3. Tumor is clinically palpable tumor
4. Symptomatic disease with facial asymmetry and cosmetic concerns
5. Diagnosis confirmed by fine needle aspiration x 2

   1. Warthin's tumor
   2. No other parotid pathologies

Exclusion Criteria:

1. Facial nerve palsy
2. History of parotid surgery
3. History or Symptoms of sialolithiasis
4. Medical facial skin conditions
5. Bleeding tendencies
6. Pregnancy
7. Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Volume reduction of Warthin's tumor compared to baseline | 1 year
  Comparison of ultrasound volumetric scan results from 45 weeks post-operative to baseline

SECONDARY OUTCOMES:
Cost and resources | 1 year
  Total cost of the procedure including all related costs
Length of in-patient stay | 1 week
  Total number of in-patient stays recorded as number of days
Operating time | 1 day
  Time required for the procedure recorded as minutes
Perioperative and post-operative complications | 1 year
  Perioperative and post-operative complications in immediate post-operatively and during the follow-up period
Cosmetic score | 1 year
  A subjective score of cosmesis graded by the patient on a scale of 1 - 4, with the higher score having worse cosmetic outcomes
Visual analogue scale for pain | 1 day
  Collected immediately post-operatively on a scale of 1 - 10, with the higher score being more painful
Visual analogue scale for patient satisfaction | 1 year
  Subjectively graded by the patient on a scale of 1-10 for outcome satisfaction, with the higher score being more satisfactory

CONTACTS AND LOCATIONS:
Overall Officials: David CM Yeung, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No